CLINICAL TRIAL: NCT02772991
Title: COmparative Prospective aNalysis betweEn Coronary angioTomography and Sensitive Troponin in Patients With Chest Pain and INtermediate Risk of Acute Coronary Syndrome in the Emergency Room - CONECTTIN Trial
Brief Title: Analysis Between Coronary Angiotomography and Sensitive Troponin in Intermediate Risk of Acute Coronary Syndrome
Acronym: CONECTTIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSInCor-TropoUS
Record Dates: First submitted 2016-04-26; First posted 2016-05-16 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2017-01

CONDITIONS: Chest Pain; Acute Coronary Syndrome
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cases (Experimental): All patients will be submmited to troponin measurements and CCTA. If CCTA shows coronary stenosis ≥ 50%, patient will initiate the ACS treatment and be hospitalized to have coronary cineangiography. If CCTA shows lesions < 50%, the patient will be discharged and monitored for 30 days. A second sampling of the troponin will be obtained from all patients three hours after the first collection in order to evaluate for an increase/decrease of troponin.
  Interventions: Other: troponin measurement

INTERVENTIONS:
Other: troponin measurement — Cardiac catheterization (for patients with >50% lesions) or discharge or in patients with intermediate risk.
  Other Names: coronary CT angiopraphy

SUMMARY:
In recent years, a large number of studies have been conducted on how to improve the treatment of patients in the Emergency Room (ER) complaining of chest pains. Great advances have been achieved recently regarding diagnostic methods aided by coronary CT angiopraphy (CCTA) and sensitive troponins. However, various questions about these methods still remain obscure and there is no effective comparison between them in patients with intermediate risk. The aim of the study is to evaluate the sensitivity and specificity of sensitivity troponins in the detection of coronary artery disease in patients with chest pain and the intermediate probability of ACS compared with CCTA.

DETAILED DESCRIPTION:
This will be a prospective and unicentric study with approximately 200 subjects recruited over a planned recruitment period of 24 months. Based on an alpha error of 0.05 and using a power of 0.8 for the primary outcomes, investigators calculated the number of individuals necessary for the study to be at least 141. All patients will be submmited to troponin measurements and CCTA. The commercial kit ADVIA Centaur® TnI-Ultra (Siemens Healthcare Diagnostics, Tarrytown, NY, USA) is used for this in automated equipment of the same brand. It is measured at the central InCor laboratory. The 99th percentile value is 0.04 ng/ml. The CCTA used will be the 320-channel Toshiba Aquilium machine. If the CCTA result shows coronary stenosis greater than or equal to 50%, the patient will initiate the ACS treatment and be hospitalized to have coronary cineangiography. In case the CCTA shows lesions of less than 50%, the patient will be discharged and monitored for 30 days by telephone. This conduct is already followed as a routine in the emergency unit at InCor for both situations. A second sampling of the troponin kit will be obtained from all patients three hours after the first collection in order to evaluate for an increase/decrease of troponin. This second troponin measurement, however, it is blinded to the main investigator, who will only have access to it after the evaluation of outcomes at the end of the study. All the data will be placed in a Microsoft Access database table and analyzed with the SAS Statview 5.0 software. The comparative analysis between the methods will be made using the area under the ROC curve and obtaining sensitivity, specificity, positive and negative predictive values, and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* chest pain for at least two hours before arriving at the emergency unit
* non-diagnostic electrocardiogram (absence of new or probable deviation of ST of at least 0.5 mV and/or T wave inversion of at least 0.2 mV)
* TIMI risk of 3 or 4
* first measurement of troponin I less than or equal to ≤ 0.03 ng/ml
* informed consent form signed.

Exclusion Criteria:

* pregnancy
* hemodynamic instability (pulmonary congestion / systolic arterial pressure lower than 90 mmHg)
* serum creatinine higher than 1.5 mg/dL
* intolerance to ß-blockers
* allergy to iodinated contrast
* asthma
* thoracic trauma within the last 30 days
* body mass index greater than 40 kg/ m2
* previous surgical myocardial revascularization
* other identified causes of troponin increase

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events according to phone contact after 30 days | 30 days
  Patients whose CCTAs show lesions with stenosis of less than 50%, compare combined outcomes (death, AMI, rehospitalization, and stroke)with the increase/decrease of troponin in the second measurement in 30 days according to phone contact.
Compare the sensitivity, specificity, and negative and positive predictive values between the high sensitivity troponin and the CCTA in the detection of an ACS. | 30 days
  ROC curve / ANOVA

SECONDARY OUTCOMES:
Stablish the cut off for troponin levels | 3 hours
  Patients whose CCTAs show coronary lesion with stenosis of more than 50%, compare with lesions with stenosis of more than 70% / acute plaque in the coronary cineangiography. In addition, compare the lesions treated in this group of patients and the increase/decrease of troponin in the second measurement; evaluate the best cut-off point regarding the percentage of variation in the troponin kit between zero and three hours that are related to the presence of lesions with stenosis of more than 70% / acute plaque in the coronary cineangiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração - HMFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No